CLINICAL TRIAL: NCT01301599
Title: Comparison Between Alpha Blocker Monotherapy and 5-alpha-reductase Inhibitor Monotherapy Following Combination Therapy in Benign Prostatic Hyperplasia
Brief Title: Comparison Between Alpha Blocker Monotherapy and 5ARI Monotherapy Following Combination Therapy in Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-09-024
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; alpha blocker; 5-alpha reductase inhibitor; combination therapy
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- combination group (Experimental): combination therapy of alpha blocker and 5-alpha-reductase inhibitor medication
  Interventions: Drug: combination therapy
- alpha blocker group (Active Comparator): alpha blocker monotherapy
  Interventions: Drug: alpha blocker monotherapy
- 5 ARI group (Active Comparator): 5 alpha-reductase inhibitor group
  Interventions: Drug: 5 alpha reductase inhibitor monotherapy

INTERVENTIONS:
Drug: combination therapy — alpha blocker and 5-alpha-reductase inhibitor medication
  Arms: combination group
Drug: alpha blocker monotherapy — alpha blocker monotherapy group
  Arms: alpha blocker group
Drug: 5 alpha reductase inhibitor monotherapy — 5 alpha reductase inhibitor monotherapy
  Arms: 5 ARI group

SUMMARY:
This study is designed to investigate the comparison between alpha blocker monotherapy and 5-alpha-reductase inhibitor monotherapy following combination therapy in benign prostatic hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 45 years old and above (with no upper limit of age)
2. patients who underwent combination therapy of alpha blocker and 5 ARI for more than 9 months
3. IPSS ≤ 12
4. Ability and willingness to correctly complete the micturition diary and questionnaire
5. Capable of understanding and having signed the informed consent form after full discussion of the research nature of the treatment and its risks and benefits

Exclusion Criteria:

1. An anticholinergic or antidiuretic if started less than 3 months prior to screening
2. Patients who had surgical treatment due to LUTS
3. Patients with suspected neurogenic bladder disorder
4. Patients with cancer of any type including cancer of the prostate or bladder
5. Patients with urethral stricture or bladder neck contracture
6. Patients with suspicious chronic prostatitis/chronic pelvic pain syndrome
7. Acute bacterial prostatitis less than 6 months prior to screening
8. Symptomatic acute urinary tract infection (UTI) less than 1 months prior to screening
9. Patients who had underwent prostatic biopsy less than one month prior to screening
10. Patients who had unstable angina or cerebral vascular disease less than 6 months prior to screening

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Numeric change of IPS and Numeric change of IPSS total score | from baseline to 12 months of treatment

SECONDARY OUTCOMES:
Changes in patients' symptom questionnaires : IPSS, ICIQ male LUTS | from baseline to 12 months of treatment
Changes in urodynamic parameters : maximal flow rate and PVR | from baseline to 12 months of treatment
change in finding of TRUS | from baseline to 12 months of treatment
Numeric Change and percent change in PSA | from baseline to 12 months of treatment
safety evaluation : incidence and severity of adverse events | 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea